CLINICAL TRIAL: NCT01066338
Title: Genome-wide Pharmacogenetic Candidate Gene SNP Array-based Approach to Predict Chemoresponse and Survival in Patients With Acute Myeloid Leukemia With Normal Karyotype
Brief Title: Genome-wide Pharmacogenetic Candidate Gene Single Nucleotide Polymorphism (SNP) Array-based Approach to Predict Chemoresponse and Survival in Patients With Acute Myeloid Leukemia With Normal Karyotype
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Dong Hwan (Dennis) Kim/Assistant professor, Samsung Medical Center
Other Study IDs: 2009-10-070
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2010-02

CONDITIONS: Myeloid Leukemia
Keywords: SNP array; prognosis; acute myeloid leukemia; normal karyotype; acute myeloid leukemia with normal karyotype
MeSH Terms: conditions — Leukemia, Myeloid; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — The stored bone marrow specimens of patients with normal karyotype AML who were treated with chemotherapy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Normal karyotype: The patients were diagnosed as acute myeloid leukemia with normal karyotype.

SUMMARY:
The most reliable prognostic marker of acute myeloid leukemia(AML) is cytogenetics by karyotyping. According to cytogenetic results, the patients with AML are classified as better, intermediate and poor prognosis groups. The normal karyotype AML was reported in about 50% of all AML and classified as intermediate risk group. However, the patients with normal karyotype AML showed various prognosis. Therefore, the further studies about subgroup analysis of normal karyotype AML are needed. Recently, the understandings of human genome polypmorphism using SNP array have been accumulated. However, the advanced researches for clinical application are not enough.

The study design is a retrospective and single-center study. The patients with normal karyotyping AML who were diagnosed from 1994 to 2008 at Samsung Medical Center (South Korea) will be enrolled. The stored bone marrow samples of enrolled patients are used for genome wide scanning by SNP array.

The purpose of present study is to develop predictive pharmacogenemic biomarkers model associated wit clinical outcomes including efficacy and toxicity in patients with AML with normal karyotype treated with chemotherapy using pharmacogenetic SNP array. And secondly, to develop enrichment clinical trial based on predictive pharmacogenomic model.

ELIGIBILITY:
Inclusion Criteria:

* patients with normal karyotype acute myeloid leukemia
* 18 years or older
* patients were treated with standard chemotherapy
* patients with available medical record and stored bone marrow specimen at time of diagnosis

Exclusion Criteria:

* no definitive criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who were diagnosed as acute myeloid leukemia with normal karyotype will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
overall response rate | within 1 month after enrollment

SECONDARY OUTCOMES:
overall survival time | within 1 month after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hwan Kim, M.D.,Ph.D., Principal Investigator — Division of Hematology and Oncology/Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea